CLINICAL TRIAL: NCT00458393
Title: Chemoprophylaxis for HIV Prevention in Men
Brief Title: Emtricitabine/Tenofovir Disoproxil Fumarate for HIV Prevention in Men
Acronym: iPrEx
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CO-US-104-0288; 10445 (Registry Identifier: DAIDS ES); 1U01AI064002 (NIH); iPrEx (Other: Study team); NCT00350324 (obsolete NCT alias)
Record Dates: First submitted 2007-04-06; First posted 2007-04-10 (Estimated); Results first posted 2018-01-24 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV; Chemoprophylaxis; Hepatitis; Viral human hepatitis; HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Hepatitis; Hepatitis, Viral, Human | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TDF/FTC (Experimental): Drug. Daily oral tablet of co-formulated 200 mg emtricitabine and 300 mg tenofovir disoproxil fumarate (TDF/FTC).
  Interventions: Drug: daily TDF/FTC
- Placebo (Placebo Comparator): Drug. Daily oral placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: daily TDF/FTC — daily oral medication
  Other Names: truvada
  Arms: TDF/FTC
Drug: Placebo — daily oral medication
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether daily use of emtricitabine/tenofovir disoproxil fumarate (FTC/TDF) can prevent HIV infection in men who also receive HIV counseling, condoms, and treatment for other sexually transmitted infections (STIs).

DETAILED DESCRIPTION:
The Joint United Nations Programme on AIDS estimates that 14,000 persons are newly infected with HIV every day worldwide; one half of these infections occur in people between the ages of 15 and 24. New infections occur despite widespread awareness of the modes of HIV transmission and the protection afforded by condom use. Effective interventions for HIV prevention are urgently needed. This study will evaluate the safety and efficacy of chemoprophylaxis for HIV prevention in men who have sex with men (MSM) who are at high risk for HIV infection despite using condoms, receiving HIV counseling, and receiving treatment for STIs, particularly hepatitis B virus (HBV) infection. A daily combination dose of emtricitabine and tenofovir disoproxil fumarate (FTC/TDF) has been selected for evaluation because it has a well-established safety record in previous studies and was demonstrated to be effective for HIV prevention in primate models. These medications have long half-lives that allow daily dosing and do not have known interactions with hormonal contraception, methadone, or tuberculosis therapies.

Once on the study drug, participants will be followed for a variable length of time, starting within 4 weeks of their screening visit and lasting up to 144 weeks. All participants will be followed for at least 8 weeks after stopping study drug. Participants who are reactive to a Hepatitis B surface antigen (HBsAg) test will be followed for hepatic flares for 16 additional weeks for a total of 24 weeks after stopping study drug. If enrolled in the optional substudy of bone mineral density, fat distribution, and fasting lipids, the participant will be asked to return for one additional visit 24 weeks after stopping study drug. Participants who HIV seroconvert during their participation will also be followed until the end of the study.

All study visits will be at 4 week intervals. At study entry, high risk, HIV uninfected MSM will be randomly assigned to receive either daily FTC/TDF or placebo, in addition to standard HIV counseling, condoms, and sexually transmitted infection (STI) management. The study will closely monitor biological and behavioral safety, including careful analysis of drug resistance, kidney and liver function, and risk behavior.

At the screening visit, participants will undergo HIV antibody and HBV testing, a medical history, a medical exam, blood and urine collection, risk behavior assessment, and STI testing. At study entry, participants will be given study medication; tested for HCV; and offered the HBV vaccine, if applicable. At all study visits, there will be HIV antibody testing, pill counts, adherence checks, study medication distribution, HIV counseling, and condom distribution. A medical history and blood will be taken on selected visits, along with STI testing and treatment if needed. Testing and treatment of STIs will be provided at no cost to the participant.

All study participants will be encouraged to join a substudy that will assess interactions between HBV infection, bone mineral density and fat distribution, and immune function. If enrolled in the substudy, the participant will be asked to return for one additional visit 24 weeks after stopping the study medication. All participants in the substudy will undergo dual energy x-ray absorptiometry (DEXA) scans, and HIV infected participants will undergo additional blood collection.

Sites will have the option of participating in the following four substudies:

The Hair Substudy: Participants who are receiving FTC/TDF will be eligible to enroll. At each 12-week follow-up study visit, hair samples will be collected and questionnaires will be completed.

The Urine Substudy: For all participants who elect to enroll in this substudy, additional testing will occur on blood and urine samples collected at each 24-week follow-up visit. An additional urine collection will occur 8 weeks after participants stop receiving FTC/TDF.

The Semen Substudy: Participants who seroconvert during the study may elect to participate in this substudy. One semen sample will be collected at participants' next study visit when plasma viral load testing is performed.

The Gonorrhea and Chlamydia Substudy: Participants in this substudy will undergo rectal and oropharyngeal swab procedures and urine collection at the 24-week study visit.

After the randomized phase ends, if the daily oral FTC/TDF arm is shown to be beneficial and safe, participants will be given the option of participating in an open label extension phase. During this extension phase, study participants will receive daily oral open-label FTC/TDF, in addition to standard counseling, condoms, and STI management.

ELIGIBILITY:
Inclusion Criteria:

* Male sex (at birth)
* HIV uninfected
* Age having reached the local age of consent
* High risk for HIV infection including any of the following: 1) No condom use during anal intercourse with a male HIV-positive partner or a male partner of unknown HIV status during the last 6 months; (2) anal intercourse with more than 3 male sex partners during the last 6 months; (3) exchange of money, gifts, shelter, or drugs for anal sex with a male partner during the last 6 months; (4) sex with a male partner and STI diagnosis during the last 6 months or at screening, or (5) sexual partner of an HIV-infected man with whom condoms are not consistently used in the last 6 months.
* Able to provide a street address of residence for themselves and one personal contact who would know their whereabouts during the study period
* Healthy enough to work, as indicated by score of 80 or greater on the Karnofsky scale
* Certain laboratory values
* A urine dipstick with a negative or trace result for both glucose and protein within 28 days of enrollment.
* Ability to understand and local language for which an informed consent form has been approved by a local IRB and registered with the study sponsor.

Inclusion Criteria for Open-Label Extension:

* Participated in a randomized, placebo-controlled, PrEP trail
* Has been unblinded
* Has provided informed consent

Exclusion Criteria:

* Previously diagnosed active and serious infections, including tuberculosis infection, osteomyelitis, or infections requiring parenteral antibiotic therapy
* Active clinically significant medical problems including heart disease (e.g., symptoms of ischemia, congestive heart failure, arrhythmia), lung disease (steroid-dependent chronic obstructive pulmonary disease), diabetes requiring hypoglycemic medication, or previously diagnosed cancer expected to require further treatment
* Acute HBV infection at the screening visit or presence of treatment indications for hepatitis B based on local practice standards; or clinical signs of hepatic cirrhosis
* History of pathological bone fractures not related to trauma
* Receiving ongoing therapy with certain HIV/AIDS-related medications or other medications as determined by the investigator
* Definitely or possibly received an anti-HIV vaccine while participating in a blinded clinical trial
* Current alcohol or drug use that, in the opinion of the investigator, may interfere with the study
* Current participation in a clinical trial or cohort study other than sub-studies of this protocol
* Any condition at enrollment that, in the opinion of the investigator, would make participation in the study unsafe or would interfere with the study
* Sites may utilize additional criteria that restrict enrollment to a subset of people who meet the protocol-defined enrollment criteria.

Exclusion Criteria for Open-Label Extension:

- Site leadership believes participant will have difficulty completing requirements

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2499 (Actual)
Dates: Start 2007-06; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert M. Grant, MD, MPH, Principal Investigator — J. David Gladstone Institutes, University of California San Francisco
Locations (11):
- United States (3):
  - San Francisco Dept. of Public Health iPrEx CRS, San Francisco, California
  - Stroger Hospital of Cook County/Core Center IPREX CRS, Chicago, Illinois
  - Fenway Community Health iPrEx CRS, Boston, Massachusetts
- Brazil (3):
  - IPEC/FIOCRUZ iPrEx CRS, Rio de Janeiro
  - Projeto Praca Onze, Universidade Federal do Rio de Janeiro iPrEx CRS, Rio de Janeiro
  - Universidade de Sao Paulo iPrEx CRS, São Paulo
- Fundación Ecuatoriana Equidad, Guayaquil, iPrEx CRS, Guayaquil, Guayas, Ecuador
- Peru (2):
  - Asociación Civil Selva Amazónica, Iquitos, iPrEx CRS, Iquitos, Maynas
  - Investigaciones Médicas en Salud (INMENSA), Lince, iPrEx CRS, Lima
- Desmond Tutu HIV Ctr. iPrEx CRS, Cape Town, South Africa
- Research Institute for Health Sciences iPrEx CRS, Chiang Mai, Thailand

REFERENCES:
- [Result] Grant RM, Lama JR, Anderson PL, McMahan V, Liu AY, Vargas L, Goicochea P, Casapia M, Guanira-Carranza JV, Ramirez-Cardich ME, Montoya-Herrera O, Fernandez T, Veloso VG, Buchbinder SP, Chariyalertsak S, Schechter M, Bekker LG, Mayer KH, Kallas EG, Amico KR, Mulligan K, Bushman LR, Hance RJ, Ganoza C, Defechereux P, Postle B, Wang F, McConnell JJ, Zheng JH, Lee J, Rooney JF, Jaffe HS, Martinez AI, Burns DN, Glidden DV; iPrEx Study Team. Preexposure chemoprophylaxis for HIV prevention in men who have sex with men. N Engl J Med. 2010 Dec 30;363(27):2587-99. doi: 10.1056/NEJMoa1011205. Epub 2010 Nov 23. PMID 21091279
- [Derived] Zivich PN, Cole SR, Edwards JK, Glidden DV, Das M, Shook-Sa BE, Shao Y, Mehrotra ML, Adimora AA, Eron JJ. HIV Prevention Among Men Who Have Sex With Men: Tenofovir Alafenamide Combination Preexposure Prophylaxis Versus Placebo. J Infect Dis. 2024 Apr 12;229(4):1123-1130. doi: 10.1093/infdis/jiad507. PMID 37969014
- [Derived] Mehrotra ML, Westreich D, McMahan VM, Glymour MM, Geng E, Grant RM, Glidden DV. Baseline Characteristics Explain Differences in Effectiveness of Randomization to Daily Oral TDF/FTC PrEP Between Transgender Women and Cisgender Men Who Have Sex With Men in the iPrEx Trial. J Acquir Immune Defic Syndr. 2019 Jul 1;81(3):e94-e98. doi: 10.1097/QAI.0000000000002037. No abstract available. PMID 31192894
- [Derived] Glidden DV, Mulligan K, McMahan V, Anderson PL, Guanira J, Chariyalertsak S, Buchbinder SP, Bekker LG, Schechter M, Grinsztejn B, Grant RM. Metabolic Effects of Preexposure Prophylaxis With Coformulated Tenofovir Disoproxil Fumarate and Emtricitabine. Clin Infect Dis. 2018 Jul 18;67(3):411-419. doi: 10.1093/cid/ciy083. PMID 29415175
- [Derived] Glidden DV, Mulligan K, McMahan V, Anderson PL, Guanira J, Chariyalertsak S, Buchbinder SP, Bekker LG, Schechter M, Grinsztejn B, Grant RM. Brief Report: Recovery of Bone Mineral Density After Discontinuation of Tenofovir-Based HIV Pre-exposure Prophylaxis. J Acquir Immune Defic Syndr. 2017 Oct 1;76(2):177-182. doi: 10.1097/QAI.0000000000001475. PMID 28639995
- [Derived] Gandhi M, Glidden DV, Mayer K, Schechter M, Buchbinder S, Grinsztejn B, Hosek S, Casapia M, Guanira J, Bekker LG, Louie A, Horng H, Benet LZ, Liu A, Grant RM. Association of age, baseline kidney function, and medication exposure with declines in creatinine clearance on pre-exposure prophylaxis: an observational cohort study. Lancet HIV. 2016 Nov;3(11):e521-e528. doi: 10.1016/S2352-3018(16)30153-9. Epub 2016 Aug 31. PMID 27658870
- [Derived] Castillo-Mancilla J, Seifert S, Campbell K, Coleman S, McAllister K, Zheng JH, Gardner EM, Liu A, Glidden DV, Grant R, Hosek S, Wilson CM, Bushman LR, MaWhinney S, Anderson PL. Emtricitabine-Triphosphate in Dried Blood Spots as a Marker of Recent Dosing. Antimicrob Agents Chemother. 2016 Oct 21;60(11):6692-6697. doi: 10.1128/AAC.01017-16. Print 2016 Nov. PMID 27572401
- [Derived] Glidden DV, Amico KR, Liu AY, Hosek SG, Anderson PL, Buchbinder SP, McMahan V, Mayer KH, David B, Schechter M, Grinsztejn B, Guanira J, Grant RM. Symptoms, Side Effects and Adherence in the iPrEx Open-Label Extension. Clin Infect Dis. 2016 May 1;62(9):1172-7. doi: 10.1093/cid/ciw022. Epub 2016 Jan 20. PMID 26797207
- [Derived] Mulligan K, Glidden DV, Anderson PL, Liu A, McMahan V, Gonzales P, Ramirez-Cardich ME, Namwongprom S, Chodacki P, de Mendonca LM, Wang F, Lama JR, Chariyalertsak S, Guanira JV, Buchbinder S, Bekker LG, Schechter M, Veloso VG, Grant RM; Preexposure Prophylaxis Initiative Study Team. Effects of Emtricitabine/Tenofovir on Bone Mineral Density in HIV-Negative Persons in a Randomized, Double-Blind, Placebo-Controlled Trial. Clin Infect Dis. 2015 Aug 15;61(4):572-80. doi: 10.1093/cid/civ324. Epub 2015 Apr 23. PMID 25908682
- [Derived] Liu A, Glidden DV, Anderson PL, Amico KR, McMahan V, Mehrotra M, Lama JR, MacRae J, Hinojosa JC, Montoya O, Veloso VG, Schechter M, Kallas EG, Chariyalerstak S, Bekker LG, Mayer K, Buchbinder S, Grant R; iPrEx Study team. Patterns and correlates of PrEP drug detection among MSM and transgender women in the Global iPrEx Study. J Acquir Immune Defic Syndr. 2014 Dec 15;67(5):528-37. doi: 10.1097/QAI.0000000000000351. PMID 25230290
- [Derived] Liegler T, Abdel-Mohsen M, Bentley LG, Atchison R, Schmidt T, Javier J, Mehrotra M, Eden C, Glidden DV, McMahan V, Anderson PL, Li P, Wong JK, Buchbinder S, Guanira JV, Grant RM; iPrEx Study Team. HIV-1 drug resistance in the iPrEx preexposure prophylaxis trial. J Infect Dis. 2014 Oct 15;210(8):1217-27. doi: 10.1093/infdis/jiu233. Epub 2014 Apr 16. PMID 24740633
- [Derived] Buchbinder SP, Glidden DV, Liu AY, McMahan V, Guanira JV, Mayer KH, Goicochea P, Grant RM. HIV pre-exposure prophylaxis in men who have sex with men and transgender women: a secondary analysis of a phase 3 randomised controlled efficacy trial. Lancet Infect Dis. 2014 Jun;14(6):468-75. doi: 10.1016/S1473-3099(14)70025-8. Epub 2014 Mar 7. PMID 24613084
- [Derived] Amico KR, Mansoor LE, Corneli A, Torjesen K, van der Straten A. Adherence support approaches in biomedical HIV prevention trials: experiences, insights and future directions from four multisite prevention trials. AIDS Behav. 2013 Jul;17(6):2143-55. doi: 10.1007/s10461-013-0429-9. PMID 23435697

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study recruited HIV uninfected participants whose sexual practices put them at risk for HIV infection. They were recruited from community clinics.
Groups:
- TDF/FTC: Daily oral emtricitabine/tenofovir disoproxil fumarate
  Emtricitabine/tenofovir disoproxil fumarate: Fixed-dose coformulation of 200 mg emtricitabine and 300 mg tenofovir disoproxil fumarate
- Placebo: Daily oral placebo
  Placebo: Placebo for emtricitabine/tenofovir disoproxil fumarate
Period: Overall Study
Arm/Group | TDF/FTC | Placebo
Started | 1251 | 1248
Completed | 942 | 953
Not Completed | 309 | 295
Not completed — Withdrawal by Subject | 67 | 80
Not completed — Physician Decision | 31 | 22
Not completed — Relocated | 77 | 81
Not completed — Lost to Follow-up | 115 | 92
Not completed — Sites marked other on the form. | 19 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TDF/FTC | Placebo | Total
Number analyzed (Participants) | 1251 | 1248 | 2499
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 92 | 101 | 193
  Between 18 and 65 years | 1158 | 1147 | 2305
  >=65 years | 1 | 0 | 1
Age, Continuous [Median (Full Range); unit: years] | 25 [18 to 67] | 24 [18 to 63] | 24 [18 to 67]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male Sex at Birth. Identify Trans | 155 | 155 | 310
  Male Sex at Birth. Identify Female | 15 | 14 | 29
  Male Sex at Birth. Identify Male | 1081 | 1079 | 2160
Region of Enrollment [Number; unit: participants]
  Ecuador | 150 | 150 | 300
  United States | 113 | 114 | 227
  Brazil | 186 | 184 | 370
  South Africa | 45 | 43 | 88
  Thailand | 57 | 57 | 114
  Peru | 700 | 700 | 1400

OUTCOME MEASURES:

1. Primary Outcome: HIV Seroconversion
Description: Confirmed HIV infection
Time Frame: Monthly follow-up through a median of 1.2 years
Population: Excludes participants who were HIV+ at enrollment (2 TDF/FTC, 8 Placebo) and those with no follow-up HIV test (25 TDF/FTC and 22 Placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | TDF/FTC | Placebo
Number analyzed (Participants) | 1224 | 1218
Participants | 48 | 83
Statistical Analysis 1: Comparison: TDF/FTC vs Placebo; Primary null hypothesis: Relative hazard of 0.7 or less. Secondary null hypothesis: Relative hazard of 1.0 or less; Test type: Superiority or Other; p = 0.002, Log Rank — secondary p-value given; stratified by site; Hazard Ratio (HR) = 0.577, 95% CI 2-sided [.404 to .824], Standard Error of Mean 0.105 — Efron correction for ties. Placebo is reference. Results typically quoted as efficacy = 100*(1-HR)

2. Primary Outcome: Grade 1 or Higher Creatinine Toxicity
Description: Creatinine which reach grade 1 (mild, 1.1 to 1.3 local upper limit of normal) or higher by the US Division of AIDS grading table (version 1) or a 50% increase in creatinine from the baseline value. The DAIDS table can be found at https://rsc.tech-res.com/docs/default-source/safety/table_for_grading_severity_of_adult_pediatric_adverse_events.pdf
Time Frame: Duration of follow-up, median 1.2 years
Population: All randomized participants which at least 1 follow-up creatinine value
Measure: Count of Participants; unit: Participants
Groups:
- TDF/FTC: Daily oral emtricitabine/tenofovir disoproxil fumarate
- Placebo: Daily oral placebo
Arm/Group | TDF/FTC | Placebo
Number analyzed (Participants) | 1216 | 1217
Participants | 32 | 24
Statistical Analysis 1: Comparison: TDF/FTC vs Placebo; Test type: Superiority; p = 0.28, Fisher Exact — p-value is not adjusted for multiple comparisons, a priori threshold for statistical significance was p < 0.05; Risk Ratio (RR) = 1.33, 95% CI 2-sided [0.79 to 2.25]; Extensive analysis and methods published in https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3966916/

3. Primary Outcome: Grade 3 or Higher Phosphorous Toxicity
Description: Grade 3 or higher phosphorous toxicity (hypophosphatemia) by the Division of AIDS Grading Table (severe, level at or below 1.9 mg/dL)
Time Frame: The entire follow-up period, median 1.2 years
Population: All participants with at least 1 follow-up phosphorus value
Measure: Count of Participants; unit: Participants
Arm/Group | TDF/FTC | Placebo
Number analyzed (Participants) | 1225 | 1226
Participants | 13 | 10
Statistical Analysis 1: Comparison: TDF/FTC vs Placebo; Test type: Superiority; p = 0.54, Fisher Exact; Risk Ratio (RR) = 1.3, 95% CI 2-sided [.57 to 2.96]

4. Primary Outcome: Grade 2, 3, or 4 Laboratory Adverse Events
Description: Number of participants with at least one Grade 2, 3, or 4 laboratory adverse events (moderate, severe of life threatening based one the US Division of AIDS Grading of adverse events, version 1.0). The table can be found at https://rsc.tech-res.com/docs/default-source/safety/table_for_grading_severity_of_adult_pediatric_adverse_events.pdf
Time Frame: Entire follow-up, median 1.2 years
Population: At participants with at least one visit with laboratory values post-baseline
Measure: Count of Participants; unit: Participants
Arm/Group | TDF/FTC | Placebo
Number analyzed (Participants) | 1229 | 1226
Participants | 70 | 79
Statistical Analysis 1: Comparison: TDF/FTC vs Placebo; Test type: Superiority; p = 0.50, Log Rank; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.65 to 1.23]

5. Primary Outcome: Grade 2, 3, or 4 Clinical Adverse Events
Description: Number of participants with at least 1 Grade 2, 3, or 4 clinical adverse events (moderate, severe of life threatening based one the US Division of AIDS Grading of adverse events, version 1.0). The table can be found at https://rsc.tech-res.com/docs/default-source/safety/table_for_grading_severity_of_adult_pediatric_adverse_events.pdf
Time Frame: Entire follow-up, median 1.2 years
Population: At participants with at least one follow-up visit
Measure: Count of Participants; unit: Participants
Arm/Group | TDF/FTC | Placebo
Number analyzed (Participants) | 1226 | 1230
Participants | 157 | 162
Statistical Analysis 1: Comparison: TDF/FTC vs Placebo; Test type: Superiority; p = 0.92, Log Rank; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.79 to 1.23]

6. Secondary Outcome: Hepatitis Flares Among Hepatitis B Virus (HBV) Infected Persons During and After Chemoprophylaxis
Description: A hepatic flare is defined as an increase in alanine transaminase or aspartate transaminase to >5 fold upper limit of normal at any visit, or an increase to >2.5 fold upper limit of normal for 3 months, within 24 weeks of permanently stopping study drug.
  More details in https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4752387/
Time Frame: Quarterly lab tests through a median follow-up of 1.2 years
Population: Those with chronic active hepatitis B at enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | TDF/FTC | Placebo
Number analyzed (Participants) | 6 | 6
Participants | 0 | 0
Statistical Analysis 1: Comparison: TDF/FTC vs Placebo; Null hypothesis of no difference; Test type: Superiority or Other; p = 1.00, Fisher Exact
Statistical Analysis 2: Comparison: TDF/FTC vs Placebo; Test type: Superiority — Desc; p = 1.00, Fisher Exact; Risk Difference (RD) = 0.00

7. Secondary Outcome: Percentage Change in Bone Mineral Density
Description: % Change from baseline in bone mineral density (100 * [(value at 24 weeks- value at baseline)/ (value at baseline)]) in in hip and L1-L4 spine by dual-energy x-ray absorptiometry
Time Frame: baseline and week 24.
Population: Participants confirmed to be HIV negative at enrollment who consented to participate in the metabolic substudy. Full details in https://www.ncbi.nlm.nih.gov/pmc/articles/pmid/25908682/
Measure: Mean (Standard Error); unit: percent change from baseline
Arm/Group | TDF/FTC | Placebo
Number analyzed (Participants) | 210 | 211
percent change from baseline
  L1-L4 Spine bone mineral density | -0.59 (0.21) | 0.32 (0.21)
  Hip bone mineral density | -0.34 (0.16) | 0.29 (0.16)
Statistical Analysis 1: Comparison: TDF/FTC vs Placebo; Test type: Superiority; p = 0.001, Mixed Models Analysis — < 0.05 for statistical significance. no adjustment for multiple comparisons; Mean Difference (Net) = -.91

8. Secondary Outcome: Percentage Change in Body Fat
Description: Percentage Change (100 * [(value at 24 weeks- value at baseline)/ (value at baseline)]) in Body Fat from Baseline by dual-energy x-ray absorptiometry
Time Frame: Baseline and Week 24
Population: All participants in the body composition substudy who made a week 24 body scan
Measure: Median (Standard Error); unit: percent change from baseline
Arm/Group | TDF/FTC | Placebo
Number analyzed (Participants) | 210 | 211
percent change from baseline | 0.0 (1.0) | 3.8 (1.0)
Statistical Analysis 1: Comparison: TDF/FTC vs Placebo; Test type: Superiority; p = 0.009, median regression; Median Difference (Net) = -3.8, 95% CI 2-sided [-6.6 to -0.95]

9. Secondary Outcome: Percentage Change in Fasting Triglycerides
Description: Percentage Change (Percentage Change (100 * [(value at 24 weeks- value at baseline)/ (value at baseline)]) in Triglycerides from Baseline from a fasting sample.
Time Frame: Baseline and Week 24
Population: All participants in the metabolic substudy with a week 24 fast triglyceride value
Measure: Median (Standard Error); unit: percent change from baseline
Arm/Group | TDF/FTC | Placebo
Number analyzed (Participants) | 199 | 194
percent change from baseline | 0.0 (3.3) | 0.0 (3.4)
Statistical Analysis 1: Comparison: TDF/FTC vs Placebo; Test type: Superiority; p = 1.00, median regression; Median Difference (Net) = 0.0, 95% CI 2-sided [-9.3 to 9.3]

10. Secondary Outcome: Percent Change in Total Cholesterol
Description: Percent change (100 * [(value at 24 weeks- value at baseline)/ (value at baseline)]) in fasting total cholesterol from baseline
Time Frame: Baseline and Week 24
Population: All participants in the metabolic substudy with a week 24 fasting cholesterol
Measure: Median (Standard Error); unit: percent change from baseline
Arm/Group | TDF/FTC | Placebo
Number analyzed (Participants) | 199 | 194
percent change from baseline | -3.2 (1.2) | -1.1 (1.2)
Statistical Analysis 1: Comparison: TDF/FTC vs Placebo; Test type: Superiority; p = 0.19, median regression; Median Difference (Net) = -2.2, 95% CI 2-sided [-5.5 to 1.1]

11. Secondary Outcome: Viral Load Among HIV Infected Participants
Description: HIV-RNA in log10 units among HIV infected participants at the time closest to HIV detection
Time Frame: At the time closest to HIV detection
Population: All HIV infections detected during the study including prior to, during and after study treatment
Measure: Mean (Standard Error); unit: log RNA copies per ml
Arm/Group | TDF/FTC | Placebo
Number analyzed (Participants) | 54 | 93
log RNA copies per ml | 5.2 (0.11) | 5.1 (0.08)
Statistical Analysis 1: Comparison: TDF/FTC vs Placebo; Test type: Superiority; p = 0.56, t-test, 2 sided; Mean Difference (Net) = 0.08, 95% CI 2-sided [-.18 to 0.33]

12. Secondary Outcome: Among HIV Infected Participants Drug Resistance
Description: Genotypic resistance by clinical assays among the seroconverters from baseline to the end of the study treatment period
Time Frame: at the time of HIV acquisition
Population: There were 2 TDF/FTC seroconversions at enrollment and 48 during follow-up. There were 8 Placebo seroconversions at enrollment and 83 during follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | TDF/FTC | Placebo
Number analyzed (Participants) | 50 | 91
Participants
  Infected at Enrollment (prior to randomization): number analyzed (Participants) | 2 | 8
  Infected at Enrollment (prior to randomization) | 2 | 1
  Infected after Randomization: number analyzed (Participants) | 48 | 83
  Infected after Randomization | 0 | 0
Statistical Analysis 1: Comparison: TDF/FTC vs Placebo; Null hypothesis is the proportion of mutations is identical; Test type: Superiority or Other; p = 1.00, Fisher Exact; Risk Ratio (RR) = 1.00; Detailed resistance data is found at https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4176446/

13. Secondary Outcome: CD4 Count Among HIV Infected Participants
Description: CD4 cell count for HIV infected participants during the trial
Time Frame: at the time infection was detected
Population: HIV infected participants during the trial including those HIV+ at baseline
Measure: Mean (95% Confidence Interval); unit: cells per cubic mm
Arm/Group | TDF/FTC | Placebo
Number analyzed (Participants) | 51 | 87
cells per cubic mm | 495 [470 to 520] | 502 [483 to 521]
Statistical Analysis 1: Comparison: TDF/FTC vs Placebo; Test type: Superiority; p = 0.32, Mixed Models Analysis; Mean Difference (Net) = -7, 95% CI 2-sided [-69 to 54]

14. Secondary Outcome: Proportion of Missed Doses by Pill Count
Description: Estimated proportion of missed doses by pill count (assuming pills taken in unreturned bottles)
Time Frame: At 24 weeks
Population: Those who bottles returned at the week 24 visit.
Measure: Mean (95% Confidence Interval); unit: proportion of pills not returned
Arm/Group | TDF/FTC | Placebo
Number analyzed (Participants) | 983 | 999
proportion of pills not returned | 0.92 [0.91 to 0.93] | 0.93 [0.92 to 0.94]
Statistical Analysis 1: Comparison: TDF/FTC vs Placebo; Null hypothesis is equal proportion of pills returned; Test type: Superiority or Other; p = 0.53, Mixed Models Analysis; Mean Difference (Net) = -0.005, 95% CI 2-sided [-0.02 to 0.01]

15. Secondary Outcome: Percentage of Missed Doses by Estimate During CASI Interview
Description: Percentage of missed doses by estimate during computer assisted structured interview
Time Frame: Week 24
Population: All participants who answered the adherence question with an estimated adherence on the week 24 computer assisted structured interview
Measure: Mean (Standard Error); unit: percentage of doses taken
Arm/Group | TDF/FTC | Placebo
Number analyzed (Participants) | 884 | 902
percentage of doses taken | 91.0 (0.5) | 91.2 (0.50)
Statistical Analysis 1: Comparison: TDF/FTC vs Placebo; Test type: Superiority; p = 0.70, t-test, 2 sided; Mean Difference (Net) = 0.25, 95% CI 2-sided [-1.1 to 1.6]; Detailed methods and results are available at https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4110718/

16. Secondary Outcome: Number of Condomless Sexual Partners With HIV Positive or Unknown Status
Description: Participants self-report of the number of sexual partners with HIV positive or unknown status in the previous 12 weeks with whom they had condomless anal sex
Time Frame: At 24 weeks
Population: Participants interviewed about sexual practices at week 24
Measure: Median (Inter-Quartile Range); unit: count
Arm/Group | TDF/FTC | Placebo
Number analyzed (Participants) | 1091 | 1114
count | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: TDF/FTC vs Placebo; Test type: Superiority; p = 0.99, Wilcoxon (Mann-Whitney) — Not adjusted for multiple comparisons and the a priori threshold for statistical significance was p < 0.05; Mean Difference (Final Values) = 0

17. Secondary Outcome: Total Number of Sexual Partners
Description: Self-reported total number of sexual partners in the previous 12 weeks.
Time Frame: 24 weeks
Population: Participants interviewed about sexual practices at week 24
Measure: Median (Inter-Quartile Range); unit: Count
Arm/Group | TDF/FTC | Placebo
Number analyzed (Participants) | 1091 | 1114
Count | 3 [1 to 6] | 3 [1 to 7]
Statistical Analysis 1: Comparison: TDF/FTC vs Placebo; Test type: Superiority; p = 0.76, Wilcoxon (Mann-Whitney) — Not adjusted for multiple comparisons, a priori threshold for statistical significance, p < 0.05; Median Difference (Final Values) = 0, 95% CI 2-sided [-.42 to .42]; Full details available in the methods section of https://www.ncbi.nlm.nih.gov/pubmed/24367497

18. Secondary Outcome: Condomless Receptive Anal Intercourse in the Previous 12 Weeks With Any Partners Regardless of Status.
Description: Self-reported condomless receptive anal intercourse in the previous 12 weeks with any partners regardless of status.
Time Frame: At 24 weeks
Population: Participants interviewed about sexual practices at week 24
Measure: Count of Participants; unit: Participants
Arm/Group | TDF/FTC | Placebo
Number analyzed (Participants) | 1091 | 1114
Participants | 332 | 348
Statistical Analysis 1: Comparison: TDF/FTC vs Placebo; Null is no difference between arms; Test type: Superiority or Other; p = 0.68, Chi-squared; Risk Difference (RD) = -0.008, 95% CI 2-sided [-0.047 to 0.030]

19. Secondary Outcome: Incidence of Confirmed Syphilis During Follow-Up
Description: Number of participants who have at least 1 confirmed syphilis infection during the study
Time Frame: All Follow-Up median of 1.2 years of follow-up
Population: Participants without active syphilis at baseline with a follow-up syphilis test.
Measure: Count of Participants; unit: Participants
Arm/Group | TDF/FTC | Placebo
Number analyzed (Participants) | 1155 | 1171
Participants | 147 | 132
Statistical Analysis 1: Comparison: TDF/FTC vs Placebo; Null hypothesis of no difference between the arms; Test type: Superiority or Other; p = 0.30, Log Rank; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.89 to 1.43]

20. Secondary Outcome: Incidence of HSV-2 During the Follow-up Period
Description: Incidence of HSV-2 during the follow-up period among those HIV-2 negative at baseline
Time Frame: Total study follow-up, a median of 1.2 years
Population: All HSV-2 negative participants with a follow-up HSV-2 test.
Measure: Count of Participants; unit: Participants
Arm/Group | TDF/FTC | Placebo
Number analyzed (Participants) | 671 | 676
Participants | 65 | 60
Statistical Analysis 1: Comparison: TDF/FTC vs Placebo; Test type: Superiority; p = 0.41, Log Rank; Hazard Ratio (HR) = 1.2, 95% CI 2-sided [0.8 to 1.7]; Details in the manuscript https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3956614/

21. Secondary Outcome: Diagnosis of Gonorrhea During the Follow-up Period
Description: Diagnosis of gonorrhea during the follow-up period by PCR
Time Frame: All of follow-up period, median of 1.2 years
Population: All participants with at least one follow-up test for gonorrhea
Measure: Count of Participants; unit: Participants
Arm/Group | TDF/FTC | Placebo
Number analyzed (Participants) | 1226 | 1229
Participants | 18 | 30
Statistical Analysis 1: Comparison: TDF/FTC vs Placebo; Test type: Superiority; p = 0.09, Log Rank; Hazard Ratio (HR) = 0.61, 95% CI 2-sided [0.34 to 1.09]

ADVERSE EVENTS:
Time Frame: Monthly follow-up with quarterly lab assessments though a median of 1.2 years of follow-up
Description: Adverse events graded by the NIH Division of AIDS grading tables, version 1.0
Arm/Group | TDF/FTC | Placebo
Serious Adverse Events (participants affected / at risk) | 92/1226 | 94/1230
Other Adverse Events (participants affected / at risk) | 906/1226 | 937/1230
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TDF/FTC (N=1226) | Placebo (N=1230)
Bone Fracture (Musculoskeletal and connective tissue disorders) | 8 (8) | 9 (9)
CREATININE INCREASE (Blood and lymphatic system disorders) | 9 (9) | 7 (7)
SUICIDE ATTEMPT (Psychiatric disorders) | 17 (17) | 14 (14)
SUICIDAL IDEATION (Psychiatric disorders) | 5 (5) | 6 (6)
ALT INCREASE (Blood and lymphatic system disorders) | 1 (1) | 4 (4)
AST (Blood and lymphatic system disorders) | 4 (4) | 5 (5)
APPENDICITIS (Hepatobiliary disorders) | 3 (3) | 3 (3)
DEPRESSION (Psychiatric disorders) | 7 (7) | 11 (11)
SUICIDAL DEPRESSION (Psychiatric disorders) | 5 (5) | 6 (6)
MAJOR DEPRESSION (Psychiatric disorders) | 5 (5) | 0 (0)
OTHER EVENTS (General disorders) | 28 (28) | 29 (29) — EVENTS AFFECTING LESS THAN A TOTAL OF 5 PARTICIPANTS
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TDF/FTC (N=1226) | Placebo (N=1230)
PHARYNGITIS (Respiratory, thoracic and mediastinal disorders) | 248 (248) | 282 (282)
PARASITIC INFECTION INTESTINAL (Gastrointestinal disorders) | 231 (231) | 216 (216)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 151 (151) | 155 (155)
BILIRUBIN INCREASE (Investigations) | 127 (127) | 132 (132)
DIARRHOEA (Gastrointestinal disorders) | 109 (109) | 123 (123)
BLOOD GLUCOSE INCREASED (Investigations) | 109 (109) | 123 (123)
BLOOD PHOSPHORUS DECREASED (Investigations) | 122 (122) | 100 (100)
HEADACHE (Nervous system disorders) | 102 (102) | 107 (107)
NASOPHARYNGITIS (Respiratory, thoracic and mediastinal disorders) | 98 (98) | 92 (92)
URETHRITIS (Renal and urinary disorders) | 84 (84) | 102 (102)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 84 (84) | 87 (87)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 76 (76) | 93 (93)
DEPRESSION (Nervous system disorders) | 81 (81) | 84 (84)
SYPHILIS (Infections and infestations) | 82 (82) | 71 (71)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 73 (73) | 76 (76)
SECONDARY SYPHILIS (Infections and infestations) | 81 (81) | 64 (64)
BLOOD AMYLASE INCREASED (Infections and infestations) | 62 (62) | 57 (57)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No